CLINICAL TRIAL: NCT03384810
Title: Causes and Outcome of Cardiac Arrest In-a University Hospital
Brief Title: Inhospital Resuscitation: Incidence, Causes and Outcome
Status: Withdrawn | Type: Observational
Why Stopped: Collecting data correctly according to the study protocol was not possible
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Associate Professor, MD, Dokuz Eylul University
Other Study IDs: 153-GOA
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: In-hospital Cardiac Arrest
Keywords: CPR; cardiac arrest; inhospital
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Define the frequency and survival pattern of cardiac arrests in relation to the hospital day of event and etiology of arrest.

DETAILED DESCRIPTION:
Define the frequency and survival pattern of cardiac arrests in relation to the hospital day of event and etiology of arrest.

The study aims to evaluate the outcome of in-hospital cardiac arrests, focusing on the relationship between etiology and outcome and, in particular, in relation to the length of hospitalization prior to the cardiac arrest. The aimed to sought to test the hypothesis that cardiac arrests occurring after longer hospitalizations were associated with lower survival rates and worse neurological outcomes compared to shorter hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Cases where the emergency help team is called

Exclusion Criteria:

* Absence of informed consent
* Lack of data records of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients who develop cardiac arrest in the hospital(Dokuz Eylul University Hospital).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
incidence of in hospital cardiac arrest | baseline
neurologic outcome of patients according to Cerebral performance category scale | until six months after return of spontaneous circulation
  The Cerebral performance category scale ranges from 1 to 5 with 1 representing intact function and 5 representing brain death.

SECONDARY OUTCOMES:
causes of intraoperative cardiac arrest among participants/patients | baseline
  Probable causes of intraoperative cardiac arrest among participants/patients Diabetes, Hypertension, Smoking, Dyslipidemia, Coronary artery disease, Chronic respiratory insufficiency, Chronic heart failure, Chronic renal insufficiency, Chronic hepatic insufficiency, Chronic neurological disease, Cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sule Ozbilgin, Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Intensive Care
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Intensive Care, Izmir, Turkey (Türkiye)